CLINICAL TRIAL: NCT03792087
Title: Efficacy & Safety of SmofKabiven Peripheral vs Compounded Emulsion: A Randomized, Active-Controlled, Open-Labelled, Multi-Centre Study in Adult Surgical Patients Requiring Parenteral Nutrition
Brief Title: Efficacy and Safety of SmofKabiven Peripheral Versus Compounded Emulsion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMKV-011-CP3
Record Dates: First submitted 2018-11-14; First posted 2019-01-03 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Parenteral Feeding; Surgery
Keywords: SmofKabiven; Nutrition; Parenteral; Abdominal surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmofKabiven Peripheral (Experimental): Continuous intravenous Infusion for SmofKabiven Peripheral via peripheral or central venous access for 14-24 hours/day. Target dose 34.3 ml per kg body weight/day. Duration of treatment 5 consecutive days.
  Interventions: Drug: SmofKabiven Peripheral
- Hospital compounded emulsion (Active Comparator): Continuous intravenous Infusion for Hospital compounded emulsion via peripheral or central venous access for 14-24 hours/day. Target dose 34.3 ml per kg body weight/day. Duration of treatment 5 consecutive days.
  Interventions: Drug: Hospital compounded emulsion

INTERVENTIONS:
Drug: SmofKabiven Peripheral — Total Parenteral Nutrition
  Other Names: Study intervention; Investigational Product
  Arms: SmofKabiven Peripheral
Drug: Hospital compounded emulsion — Total Parenteral Nutrition
  Other Names: Control; Comparator
  Arms: Hospital compounded emulsion

SUMMARY:
The present protocol describes a randomized, open-labelled study in which either SmofKabiven Peripheral or a hospital compounded control Parenteral Nutrition (PN) regimen will be given to adult surgical patients for 5 consecutive days.

As serum prealbumin is a well-established surrogate efficacy parameter reflecting the patient´s nutritional status, the absolute change of the serum prealbumin level at the day of the final study visit compared to baseline will represent the primary efficacy parameter in the present study.

DETAILED DESCRIPTION:
In addition, other variables will be assessed in this study, i.e., C-reactive Protein (CRP), free fatty acids, immunology parameters, taurine, comparison of the time required for Total Parenteral Nutrition (TPN) preparation of the two groups, the results of physical examination, vital signs, relevant nutrition- and safety-related laboratory parameters in venous blood and urine, the results of an Electrocardiography (ECG), and the number, severity, seriousness, clinical relevance, relatedness and outcome of Adverse Events (AEs). The aim of the planned study is to demonstrate that SmofKabiven Peripheral is not inferior to the comparative drug (compounded emulsion).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is scheduled to undergo elective abdominal surgery
2. Female or male patient, age between 18 and 75 years (inclusively)
3. Postoperatively, patient is expected to receive 100% of the total daily energy demand via PN for at least 5 consecutive days
4. Body Mass Index (BMI) ≥ 16 and ≤ 30 kg /m2, and actual body weight ≥ 40 kg
5. Patient is capable to give Informed Consent, agrees to participate in the study, and signs the Informed Consent Form

Exclusion Criteria:

1. Patient has received PN or parenteral amino acids in the last 10 days before randomization (exception: administration of glucose will be allowed)
2. Severe liver insufficiency or AST, ALT or total bilirubin at least 1.5-times higher than the upper limit of normal range
3. International Normalised Ratio (INR) at least 1.5 times higher than the upper limit of normal range
4. Uncontrolled hyperglycaemia, fasting blood glucose > 180 mg/ dl (10 mmol/L)
5. Severe renal impairment defined as serum creatinine value at least 1.5 times higher than the upper limit of normal range
6. Serious hyperlipidaemia (serum cholesterol and/or triglycerides and/or LDL-C level at least 1.5 times higher than the upper limit of normal range)
7. Inborn abnormality of amino acid metabolism
8. Present signs of acute pancreatitis, hypothyroidism or hyper-thyroidism as diagnosed clinically
9. Serum level of any of the electrolytes (sodium, potassium, magnesium, total calcium, chloride, phosphate) above the upper limit of the normal range
10. Known unstable metabolism (e.g., known metabolic acidosis)
11. Known hypersensitivity to fish-, egg-, soybean, or peanut protein or to any of the active substances or excipients of the study drugs
12. General contraindications to infusion therapy: acute pulmonary oedema, hyperhydration, and decompensated cardiac insufficiency /congestive heart failure
13. Unstable conditions (e.g., acute myocardial infarction, stroke, embolism, severe sepsis, shock)
14. Drug abuse and/or chronic alcoholism
15. Psychiatric diseases, epilepsy
16. Administration of growth hormones within the previous 4 weeks before surgery, or chronic maintenance therapy with systemic glucocorticoids 4 weeks before surgery
17. Participation in a clinical study with an investigational drug or an investigational medical device within one month prior to start of study or during study
18. Patient is pregnant or lactating and intends to continue breast-feeding
19. Development of intraoperative/ postoperative conditions (assessed after surgery and before enrollment of patients):

    1. Intra-operative blood loss > 1000ml;
    2. Development of a condition in which PN is contraindicated;
    3. Intra- or postoperative urine output <0.5 ml/kg/h;
    4. Need for postoperative haemo-filtration or dialysis;
    5. Contraindication or inability to obtain peripheral or central venous catheter access;
    6. Intra-operative decision on limited treatment, e.g. due to diagnosis of carcinomatosis;
    7. Intra-operative severe complications including resuscitation, hemorrhagic and septic shock, acute single and multiple organ dysfunction including pulmonary, hepatic, and renal dysfunction prohibiting early postsurgical extubation, requiring liver-specific treatment and renal replacement therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Serum Prealbumin | 6 days
  Change in Serum Prealbumin

SECONDARY OUTCOMES:
C-reactive Protein (CRP) | 6 days
  Change in CRP
Linoleic acid | 6 days
  Change in linoleic acid
Linolenic acid | 6 days
  Change in linolenic acid
Arachidonic acid | 6 days
  Change in arachidonic acid
Eicosapentaenoic acid (EPA) | 6 days
  Change in EPA
Docosahexaenoic acis (DHA) | 6 days
  Change in DHA
Thromboxane B3 (TXB3) | 6 days
  Change in TXB3
Thromboxane B2 (TXB2) | 6 days
  Change in TXB2
Interleukin (IL)-1 | 6 days
  Change in IL-1
IL-2 | 6 days
  Change in IL-2
IL-6 | 6 days
  Change in IL-6
Cluster of Differentiation 4 (CD4) /Cluster of Differentiation 8 (CD8) | 6 days
  Change in CD4/CD8
Plasma amino acid (taurine) | 6 days
  Change in plasma amino acid (taurine)

OTHER OUTCOMES:
Adverse Events (AE) | up to 16 days
  Coded according to Medical Dictionary for Regulatory Affairs (MedDRA) by System Organ Class (SOC) and preferred term
Local intolerance for peripherally infusion | 6 days
  Reported as AE
Development of phlebitis | 6 days
  Reported as AE
Development of thrombophlebitis | 6 days
  Reported as AE
Blood pressure | up to 16 days
  Vital signs
Heart rate | up to 16 days
  Vital signs
Respiratory rate | up to 16 days
  Vital signs
Body temperature | up to 16 days
  Vital signs
Physical examination | up to 16 days
  Examination of abnormal findings in any system/organ
Red blood cell (RBC) count | up to 16 days
  Laboratory variables
Total white blood cell (WBC) count | up to 16 days
  Laboratory variables
Haemoglobin (Hb) | up to 16 days
  Laboratory variables
Haematocrit (Hct) | up to 16 days
  Laboratory variables
Platelets | up to 16 days
  Laboratory variables
Creatinine | up to 16 days
  Laboratory variables
Urea | up to 16 days
  Laboratory variables
Sodium | up to 16 days
  Laboratory variables
Potassium | up to 16 days
  Laboratory variables
Magnesium | up to 16 days
  Laboratory variables
Total calcium | up to 16 days
  Laboratory variables
Chloride | up to 16 days
  Laboratory variables
Phosphate | up to 16 days
  Laboratory variables
Aspartate aminotransferase (AST) | up to 16 days
  Laboratory variables
Alanine aminotransferase (ALT) | up to 16 days
  Laboratory variables
Alkaline phosphatase (AP) | up to 16 days
  Laboratory variables
Gamma-glutamyl transpeptidase (γ-GT) | up to 16 days
  Laboratory variables
Lactate dehydrogenase (LDH) | up to 16 days
  Laboratory variables
Total and direct bilirubin | up to 16 days
  Laboratory variables
Albumin | up to 16 days
  Laboratory variables
Total protein | up to 16 days
  Laboratory variables
Glucose | up to 16 days
  Laboratory variables
Cholesterol | up to 16 days
  Laboratory variables
Triglycerides | up to 16 days
  Laboratory variables
Low Density Lipoprotein (LDL)-C | up to 16 days
  Laboratory variables
High Density Lipoprotein (HDL)-C | up to 16 days
  Laboratory variables
Fibrinogen | up to 16 days
  Laboratory variables
Activated partial thromboplastin time (APTT) | up to 16 days
  Laboratory variables
Prothrombin time (PT) | up to 16 days
  Laboratory variables
International Normalised Ratio (INR) | up to 16 days
  Laboratory variables
power of hydrogen (pH) value | up to 16 days
  Urine analysis
Bilirubin | up to 16 days
  Urine analysis
Protein | up to 16 days
  Urine analysis
WBC | up to 16 days
  Urine analysis
RBC | up to 16 days
  Urine analysis
Urine Glucose | up to 16 days
  Urine analysis
Ketone body | up to 16 days
  Urine analysis
ECG | up to 16 days
  Electrocardiogram to assess cardiac disorders (e.g. Myocardial infarction, Pericarditis, QT interval Prolongation, etc.)
Preparation time | 5 days
  Comparison of the time required for TPN preparation for the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Wu Guohao, MD, Principal Investigator — Fudan University
Locations (5):
- China (5):
  - Beijing Friendship Hospital Capital Medical University, Beijing
  - Peking University People's Hospital, Beijing
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Zhongshan Hospital, Fudan University, Shanghai

REFERENCES:
- [Background] Calder PC. n-3 fatty acids, inflammation, and immunity--relevance to postsurgical and critically ill patients. Lipids. 2004 Dec;39(12):1147-61. doi: 10.1007/s11745-004-1342-z. PMID 15736910
- [Background] Mayer K, Gokorsch S, Fegbeutel C, Hattar K, Rosseau S, Walmrath D, Seeger W, Grimminger F. Parenteral nutrition with fish oil modulates cytokine response in patients with sepsis. Am J Respir Crit Care Med. 2003 May 15;167(10):1321-8. doi: 10.1164/rccm.200207-674OC. Epub 2003 Feb 25. PMID 12615625
- [Background] Novak TE, Babcock TA, Jho DH, Helton WS, Espat NJ. NF-kappa B inhibition by omega -3 fatty acids modulates LPS-stimulated macrophage TNF-alpha transcription. Am J Physiol Lung Cell Mol Physiol. 2003 Jan;284(1):L84-9. doi: 10.1152/ajplung.00077.2002. Epub 2002 Aug 30. PMID 12388359
- [Background] Pluess TT, Hayoz D, Berger MM, Tappy L, Revelly JP, Michaeli B, Carpentier YA, Chiolero RL. Intravenous fish oil blunts the physiological response to endotoxin in healthy subjects. Intensive Care Med. 2007 May;33(5):789-797. doi: 10.1007/s00134-007-0591-5. Epub 2007 Mar 22. PMID 17377770
- [Background] Xiong J, Zhu S, Zhou Y, Wu H, Wang C. Regulation of omega-3 fish oil emulsion on the SIRS during the initial stage of severe acute pancreatitis. J Huazhong Univ Sci Technolog Med Sci. 2009 Feb;29(1):35-8. doi: 10.1007/s11596-009-0107-3. Epub 2009 Feb 18. PMID 19224159
- [Background] Helmut Grimm, A balanced lipid emulsion-A new concept in parenteral nutrition. Clinical Nutrition Supplements (2005) 1, 25-30.
- [Background] Grimm H, Mertes N, Goeters C, Schlotzer E, Mayer K, Grimminger F, Furst P. Improved fatty acid and leukotriene pattern with a novel lipid emulsion in surgical patients. Eur J Nutr. 2006 Feb;45(1):55-60. doi: 10.1007/s00394-005-0573-8. Epub 2005 Jul 22. PMID 16041475
- [Background] Puder M, Valim C, Meisel JA, Le HD, de Meijer VE, Robinson EM, Zhou J, Duggan C, Gura KM. Parenteral fish oil improves outcomes in patients with parenteral nutrition-associated liver injury. Ann Surg. 2009 Sep;250(3):395-402. doi: 10.1097/SLA.0b013e3181b36657. PMID 19661785
- [Background] Gura KM, Duggan CP, Collier SB, Jennings RW, Folkman J, Bistrian BR, Puder M. Reversal of parenteral nutrition-associated liver disease in two infants with short bowel syndrome using parenteral fish oil: implications for future management. Pediatrics. 2006 Jul;118(1):e197-201. doi: 10.1542/peds.2005-2662. PMID 16818533
- [Background] Alwayn IP, Gura K, Nose V, Zausche B, Javid P, Garza J, Verbesey J, Voss S, Ollero M, Andersson C, Bistrian B, Folkman J, Puder M. Omega-3 fatty acid supplementation prevents hepatic steatosis in a murine model of nonalcoholic fatty liver disease. Pediatr Res. 2005 Mar;57(3):445-52. doi: 10.1203/01.PDR.0000153672.43030.75. Epub 2005 Jan 19. PMID 15659701
- [Background] Bouletreau P, Chassard D, Allaouchiche B, Dumont JC, Auboyer C, Bertin-Maghit M, Bricard H, Ecochard R, Rangaraj J, Chambrier C, Schneid C, Cynober L. Glucose-lipid ratio is a determinant of nitrogen balance during total parenteral nutrition in critically ill patients: a prospective, randomized, multicenter blind trial with an intention-to-treat analysis. Intensive Care Med. 2005 Oct;31(10):1394-400. doi: 10.1007/s00134-005-2771-5. Epub 2005 Aug 24. PMID 16132885
- [Background] Sergi G, Coin A, Enzi G, Volpato S, Inelmen EM, Buttarello M, Peloso M, Mulone S, Marin S, Bonometto P. Role of visceral proteins in detecting malnutrition in the elderly. Eur J Clin Nutr. 2006 Feb;60(2):203-9. doi: 10.1038/sj.ejcn.1602289. PMID 16234837
- [Background] Shenkin A. Serum prealbumin: Is it a marker of nutritional status or of risk of malnutrition? Clin Chem. 2006 Dec;52(12):2177-9. doi: 10.1373/clinchem.2006.077412. No abstract available. PMID 17138848
- [Background] Young GA, Hill GL. Assessment of protein-calorie malnutrition in surgical patients from plasma proteins and anthropometric measurements. Am J Clin Nutr. 1978 Mar;31(3):429-35. doi: 10.1093/ajcn/31.3.429. PMID 415592
- [Background] Young GA, Collins JP, Hill GL. Plasma proteins in patients receiving intravenous amino acids or intravenous hyperalimentation after major surgery. Am J Clin Nutr. 1979 Jun;32(6):1192-9. doi: 10.1093/ajcn/32.6.1192. PMID 87126
- [Background] Young GA, Hill GL. A controlled study of protein-sparing therapy after excision of the rectum: effects of intravenous amino acids and hyperalimentation on body composition and plasma amino acids. Ann Surg. 1980 Aug;192(2):183-91. doi: 10.1097/00000658-198008000-00009. PMID 6773484
- [Background] Chinese medical clinical guidelines parenteral enteral nutrition 2008, edited by Chinese Medical Association, People's Medical Publishing House.
- [Background] Bernstein LH. The systemic inflammatory response syndrome C-reactive protein and transthyretin conundrum. Clin Chem Lab Med. 2007;45(11):1566-7; author reply 1568-9. doi: 10.1515/CCLM.2007.334. No abstract available. PMID 17970714
- [Background] SSPC. Intralipid 20%, Summary of Product Characteristics, dated 14 February 2007
- [Background] SSPC. Novamin 11.4%, Summary of Product Characteristics, dated 01 December 2013
- [Background] McClave SA, Martindale RG, Vanek VW, McCarthy M, Roberts P, Taylor B, Ochoa JB, Napolitano L, Cresci G; A.S.P.E.N. Board of Directors; American College of Critical Care Medicine; Society of Critical Care Medicine. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2009 May-Jun;33(3):277-316. doi: 10.1177/0148607109335234. No abstract available. PMID 19398613
- [Background] Braga M, Ljungqvist O, Soeters P, Fearon K, Weimann A, Bozzetti F; ESPEN. ESPEN Guidelines on Parenteral Nutrition: surgery. Clin Nutr. 2009 Aug;28(4):378-86. doi: 10.1016/j.clnu.2009.04.002. Epub 2009 May 21. PMID 19464088
- [Background] Chowdary KV, Reddy PN. Parenteral nutrition: Revisited. Indian J Anaesth. 2010 Mar;54(2):95-103. doi: 10.4103/0019-5049.63637. PMID 20661345
- [Background] Singer P, Berger MM, Van den Berghe G, Biolo G, Calder P, Forbes A, Griffiths R, Kreyman G, Leverve X, Pichard C, ESPEN. ESPEN Guidelines on Parenteral Nutrition: intensive care. Clin Nutr. 2009 Aug;28(4):387-400. doi: 10.1016/j.clnu.2009.04.024. Epub 2009 Jun 7. PMID 19505748
- [Background] Fresenius Kabi. SomfKabiven Peripheral, emulsion for infusion. Summary of Product Characteristics, dated September.29. 2009